CLINICAL TRIAL: NCT03399669
Title: The Continuation of Gefitinib Treatment Beyond Progression in Non-small Cell Lung Cancer Patients With EGFR Mutation: A Phase II Single Arm Prospective Study
Brief Title: The Continuation of Gefitinib Treatment Beyond Progression in Non-small Cell Lung Cancer Patients With EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, MD,PhD,Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-11-095
Record Dates: First submitted 2018-01-09; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gefitinib (Experimental): Patients will be treated 250 mg/day of gefitinib orally (1 cycle for 28 days). Cycles were repeated until disease progression, unacceptable toxicity, or until the patient or the investigator requested therapy discontinuation.
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib — Patients will be treated 250 mg/day of gefitinib orally (1 cycle for 28 days). Cycles were repeated until disease progression, unacceptable toxicity, or until the patient or the investigator requested therapy discontinuation.

SUMMARY:
Although EGFR-TKIs such as gefitinib, erlotinib or afatinib are recommended as first-line therapy in patients with advanced, recurrent or metastatic nonsquamous NSCLC patients who have known active EGFR mutation and achieved response to EGFR TKIs experience disease progression eventually with 10-14 moths of median progression free survival.6 Platinum-doublets combination chemotherapy remains standard of care for patients with progressive disease. However, patients may derive benefit from EGFR TKIs after RECIST-assessed progression especially for those who experience slow progression. And previous report suggested that premature discontinuation of EGFR TKIs has resulted in rapid progression in symptoms and tumor growth.7 Recently, a prospective phase II single arm study in Asian patients with EGFR mutation-positive NSCLC to determine the continuation of erlotinib beyond progression judged by investigators showed that additional PFS of 3.1 months can be achieved with continuation of erlotinib without serious additional toxicities.8 Until now, no prospective study has been conducted for gefitinib.

In this study the continuation of gefitinib beyond RECIST progression will be investigated to determine the clinical outcomes including the duration of treatment and safety.

This is a single-arm phase II trial to evaluate the efficacy and safety of continuation of gefitinib in EGFR mutant NSCLC patients who experience RECIST progression. Based on the results of "ASPIRATION" study, the median PFS for continuation of gefitinib will be around 3 months. The study treatment will be of no interest if the true median PFS is 2.5 months or shorter. In contrast, it will be of interest if the true median PFS is 3.5 months or longer. Considering 1 sided alpha of 0.05 and 90% of power, 95 patients are required. A total of 100 patients will be needed considering 5% of drop-out rate. 6 months of accrual and additional 6 months of follow-up will be assumed for this study.

Patients will be treated 250 mg/day of gefitinib orally (1 cycle for 28 days). Cycles were repeated until disease progression, unacceptable toxicity, or until the patient or the investigator requested therapy discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIB/IV or recurrent NSCLC with activating EGFR mutation in exon 18 through exon 21 except T790M
* Patients who achieved complete/partial response more than 4 months or stable disease more than 6 months with first-line or second line gefitinib
* Patients who experience disease progression by RECIST 1.1 criteria
* Age ≥ 18years
* ECOG performance status of 0 to 2
* Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; total bilirubin ≤1.5 UNL; AST and/or ALT < 5 UNL, CCr ≥ 50mL/min
* Baseline adverse event of gefitinib ≤ Grade 2
* Written informed consent form

Exclusion Criteria:

* Prior treatment with EGFR TKI
* Patients who required dose reduction of gefitinib
* Surgery undertaken less than 4 weeks before the study
* Localized radiotherapy unless completed more than 2 weeks before the study
* Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
* Pregnant or nursing women ( Women of reproductive potential have to agree to use an effective contraceptive method (hormonal or barrier methods))
* Uncontrolled symptomatic brain metastasis
* Prior history of malignancy within 5 years from study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, well-treated thyroid cancer
* Concomitant use of CYP3A4 inducers/inhibitors
* Prolonged QT interval in ECG (QTc >450 msec)
* Patients who cannot take a medicine orally or who have a gastrointestinal absorption disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2015-02-17 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from RECIST progression to secondary disease progression | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided